CLINICAL TRIAL: NCT03615768
Title: A Multi-center, Randomized, Single-blind, Paralelle, Positive Controlled Phase III Study to Evaluate the Efficacy and Safety of Adapalene-Clindamycin Combination Gel in the Treatment of Moderate Acne Vulgaris
Brief Title: A Study to Evaluate the Efficacy and Safety of Adapalene-Clindamycin Combination Gel in the Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Collaborators: Zhaoke (Guangzhou) Ophthalmology Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZK-ACG-201712
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene; Clindamycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adapalene-Clindamycin Combination Gel (Experimental)
  Interventions: Combination Product: Adapalene-Clindamycin Combination Gel
- Adapalene Gel (Active Comparator)
  Interventions: Drug: Adapalene Gel
- Clindamycin Gel (Active Comparator)
  Interventions: Drug: Clindamycin Gel

INTERVENTIONS:
Combination Product: Adapalene-Clindamycin Combination Gel — 5mg Adapalene/50mg Clindamycin per 5g, applied nightly for 12 weeks
  Arms: Adapalene-Clindamycin Combination Gel
Drug: Adapalene Gel — Differin 0.1% Gel, applied nightly for 12 weeks
  Other Names: Differin
  Arms: Adapalene Gel
Drug: Clindamycin Gel — Clindamycin Phosphate 1% Gel applied twice daily for 12 weeks
  Other Names: Clindamycin
  Arms: Clindamycin Gel

SUMMARY:
This is a study to see if Adapalene-Clindamycin Combination Gel is effective and safe in the treatment of acne vulgaris, compared to adapalene gel alone and clindamycin gel alone. Adapalene and clindamycin have been reported to have a better effect in acne treatment when used together. This new formulation is also easier to use as it combines two products into a single gel and only needs to be used once a day.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 12-40 years old
* Diagnosis of Grade II-III acne vulgaris with Pillsbury grading system
* Provide written informed consent if the subject is aged 18 or older. Ages 12-17 should provide written assent and written informed consent from patient's parent or legal guardian.

Exclusion Criteria:

* Known hypersensitivity to adapalene, clindamycin hydrochloride, clindamycin phosphate, lincomycin or any ingredient of the study drug, or of allergic constitution
* Secondary Acne, such as occupational acne and steroid acne
* Has a dermatological condition of the face that could interfere with the clinical evaluations, such as sunburn, psoriasis, seborrheic dermatitis or eczema
* History of Crohn's disease, ulcerative colitis or antibiotic-associated colitis
* History of serious heart disease or hypertension
* Serious liver or kidney disease, AST or ALT more than twice the upper limit of normal, or Cr above normal
* Serious endocrine, hematologic or psychiatric disease
* Known immunocompromised conditions, or require long-term steroids or immunosuppressants
* Females who are pregnant, lactating, or not willing to use effective contraception
* Drug or alcohol abuse
* Used any topical acne treatment within 2 weeks
* Used any systemic retinoid, antibiotic or other acne treatment
* Used any investigational drugs or device within 3 months, or concurrently enrolled in another clinical trial
* Patient who the investigator deemed to be unsuitable for any reason

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1617 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-04-07 (Actual)

PRIMARY OUTCOMES:
Percentage Change From Baseline in Total Lesion Counts | Week 12
  Percent change from Baseline in total lesions counts in each treatment group at Week 12.
Proportion of patients who has at least a two-point reduction in Investigator Global Assessment (IGA) compared to baseline | Week 12

SECONDARY OUTCOMES:
Percentage change from baseline in inflammatory lesion counts | Week 12
  Percent change from baseline in inflammatory lesions count in each treatment group at Week 12.
Percentage change from baseline in non-inflammatory lesion counts | Week 12
  Percent change from baseline in non-inflammatory lesions count in each treatment group at Week 12.
Change from baseline in inflammatory lesion counts | Week 12
  Absolute change from baseline in inflammatory lesion counts in each treatment group at Week 12.
Change from baseline in non-inflammatory lesion counts | Week 12
  Absolute change from baseline in non-inflammatory lesion counts in each treatment group at Week 12.
Change from baseline in total lesion counts | Week 12
  Absolute change from baseline in total lesions counts in each treatment group at Week 12.
Change from baseline in Investigator's Global Assessment (IGA) | Week 12
  Absolute change from baseline in Investigator's Global Assessment (IGA) in each treatment group at Week 12.
Treatment success rate | Week 12
  The proportion of subjects in each treatment group achieving "success" at Week 12, with "success" defined as an IGA score of "clear (score=0)" or "almost clear (score=1)"; if IGA score at baseline is 2, success is only achieved if IGA score is 0 at Week 12.

OTHER OUTCOMES:
Local Adverse Reactions | Week 2, Week 4, Week 8 and Week 12
  Local Adverse Reactions including erythema, scaling, stinging, burning and pruritus scored by severity

CONTACTS AND LOCATIONS:
Overall Officials: Heng Gu, MD, Principal Investigator — Institute of Dermatology and Hospital for Skin Diseases, Chinese Academy of Medical Sciences
Locations (1):
- Institute of Dermatology and Hospital for Skin Diseases, Chinese Academy of Medical Sciences, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luan C, Yang WL, Yin JW, Deng LH, Chen B, Liu HW, Zhang SM, Han J, Liu ZJ, Dai XR, Yin QJ, Yu XH, Chen K, Gu H, Li BXY. Efficacy and Safety of a Fixed-Dose Combination Gel with Adapalene 0.1% and Clindamycin 1% for the Treatment of Acne Vulgaris (CACTUS): A Randomized, Controlled, Assessor-Blind, Phase III Clinical Trial. Dermatol Ther (Heidelb). 2024 Nov;14(11):3097-3112. doi: 10.1007/s13555-024-01286-x. Epub 2024 Nov 1. PMID 39487326